CLINICAL TRIAL: NCT07284524
Title: The Dynamic Dual-Mode Alignment Optimization and Intelligent Precision Knee Preservation System for Knee Osteoarthritis
Brief Title: Intelligent Precision Knee Preservation System for Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025-307
Record Dates: First submitted 2025-09-07; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis (Knee OA)
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MA group (Placebo Comparator): HTO utilizing osteotomy-specific plates (e.g., TOMOFIX), targeting the mechanical (Fujisawa) alignment (MA).
  Interventions: Behavioral: HTO procedure
- KA Group (Experimental): HTO utilizing osteotomy-specific plates (e.g., TOMOFIX), targeting a kinematic alignment (KA) target
  Interventions: Behavioral: HTO procedure
- DA group (Experimental): HTO utilizing osteotomy-specific plates (e.g., TOMOFIX), targeting with dynamic dual-mode alignment (DA) optimization combined with the intelligent precision knee-preserving system
  Interventions: Behavioral: HTO procedure

INTERVENTIONS:
Behavioral: HTO procedure — HTO procedure for knee osteoarthritis

SUMMARY:
The goal of this clinical trial is to verify whether the "dynamic dual-mode alignment optimization + intelligent precision knee-preserving system" (integrating static/kinematic target alignment, CT-based preoperative three-dimensional [3D] planning, 3D-printed guide plates, and intraoperative augmented reality [AR] real-time feedback) achieves a greater relative reduction in peak knee adduction moment (KAM) at 12 months postoperatively, while maintaining or improving knee clinical function and without increasing perioperative or long-term complication rates, compared with traditional knee-preserving strategies. The target population is patients aged 40-70 years with knee osteoarthritis (KOA; Kellgren-Lawrence grade II-III) who require high tibial osteotomy (HTO) for unilateral medial-compartment disease with mild-to-moderate varus deformity and who meet the inclusion and exclusion criteria.

The main questions are:

* Can the dynamic dual-mode alignment + intelligent precision system achieve a greater relative reduction in peak KAM at 12 months postoperatively than traditional knee-preserving strategies?
* Can this system improve static alignment accuracy, dynamic load parameters (e.g., KAM impulse and varus thrust), and patient-reported outcome (PRO) scores without increasing complication rates?
* Can 3D-printed patient-specific instrumentation (PSI) guide plates and real-time AR feedback reduce intraoperative radiation exposure and shorten operative time compared with traditional methods?

Researchers will compare:

Kinematic alignment (KA), traditional mechanical alignment (MA), and dynamic dual-mode alignment (DA) to evaluate the relative performance of alignment strategies;

3D-printed PSI-guided HTO versus traditional fluoroscopy-guided HTO to assess the efficacy of PSI; and

AR-assisted intraoperative adjustment versus traditional fluoroscopy-based adjustment to evaluate the precision of AR navigation.

Participants will:

* Complete preoperative assessments, including laboratory tests (complete blood count, biochemistry, coagulation), imaging (full-length, weight-bearing lower-limb radiographs; knee CT and/or MRI as indicated), 3D gait analysis (to measure KAM, KAM impulse, and varus thrust), and PRO assessments (KOOS, WOMAC, and Lysholm scores)
* Receive assigned surgical interventions: the DA group will undergo HTO guided by dual-mode alignment plus 3D-printed PSI and intraoperative AR feedback; the MA and KA groups will undergo HTO based on traditional or kinematic alignment, respectively; the traditional HTO group will undergo surgery relying on intraoperative fluoroscopy and surgeon experience.
* Attend follow-up visits at 6 weeks, 3 months, 6 months, and 12 months postoperatively, including imaging to assess alignment accuracy and bone healing, gait analysis, PRO assessments, and complication monitoring.
* Record medication use and rehabilitation compliance throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 70 years;
2. Unilateral medial compartment knee osteoarthritis (mild to moderate pain);
3. Mild to moderate varus deformity (5°-15°);
4. Coronal MRI showing medial meniscus extrusion (MME) >3 mm and flexion contracture <10°;
5. Intact lateral meniscus and articular cartilage;

Exclusion Criteria:

1. Patients with concomitant inflammatory arthritis (e.g., rheumatoid arthritis) or systemic inflammatory diseases;
2. Patients with severe varus deformity (>10°) or flexion contracture >10°;
3. Patients with lateral meniscus pathology (tear, discoid meniscus) or knee joint instability;
4. Patients with a history of major knee trauma, infection, or prior knee surgery;
5. Patients with severe patellofemoral osteoarthritis;
6. Patients with advanced medial compartment osteoarthritis (bone-on-bone contact or knee subluxation);
7. Patients who refuse second-look arthroscopy or participation in the study;
8. Patients unable to complete at least 12 months of follow-up;
9. Patients with severe osteoporosis;
10. Patients with cognitive impairment.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Relative ΔKAM (%) | Preoperative, and 6 weeks, 3 months, 6 months, 12 months postoperatively
  Relative ΔKAM (%) = [(KAM_follow-up - KAM_preoperative) / KAM_preoperative] × 100%
HKA Accuracy | Preoperative, and 12 months postoperatively
  HKA accuracy is defined as the proportion of operated knees whose hip-knee-ankle (HKA) angle falls within the prespecified target window (±2°) on full-length, weight-bearing radiographs at 12 months postoperatively.
KOOS score | Preoperative, and 6 weeks, 3 months, 6 months, 12 months postoperatively
  Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-administered questionnaire (paper or electronic; 1-week recall) with 42 items across five subscales: Symptoms, Pain, Activities of Daily Living (ADL), Sport and Recreation Function (Sport/Rec), and Knee-related Quality of Life (QOL). Items are rated 0-4. For each subscale, raw scores are summed and transformed to a 0-100 scale using:
  Score = 100 - [(sum of item scores × 100) ÷ (4 × number of items)]. Minimum = 0 (worst outcome); Maximum = 100 (best outcome); higher scores indicate better status.
  Subscales are reported separately. If reported, "KOOS4" is the mean of Pain, Symptoms, Sport/Rec, and QOL, also on a 0-100 scale with 0 = worst and 100 = best (higher = better).
WOMAC Osteoarthritis Index | Preoperative, and 6 weeks, 3 months, 6 months, 12 months postoperatively
  The Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index is a self-administered questionnaire designed to assess pain, stiffness, and physical function in patients with hip and knee osteoarthritis. It contains 24 items across three subscales: pain (5 items), stiffness (2 items), and physical function (17 items). Each item is scored on a Likert scale (0-4; none to extreme) or sometimes a 100-mm visual analogue scale, depending on the version used. Scores are summed for each subscale and can be normalized to a 0-100 scale (higher scores indicate worse symptoms).
HSS score | Preoperative, and 6 weeks, 3 months, 6 months, 12 months postoperatively
  The Hospital for Special Surgery (HSS) score is a clinician-administered questionnaire designed to evaluate knee function. It includes six domains: pain (30 points), function (22 points), range of motion (18 points), muscle strength (10 points), flexion deformity (10 points), and instability (10 points), with deductions for the use of walking aids. The maximum score is 100 points, with higher scores indicating better knee function: >85 excellent, 70-84 good, 60-69 fair, and <60 poor.
Lysholm score | Preoperative, and 6 weeks, 3 months, 6 months, 12 months postoperatively
  The Lysholm score is a patient-reported outcome measure originally designed for knee ligament injuries, widely used to evaluate knee symptoms and function. It consists of 8 items: limp, need for support, locking, instability, pain, swelling, stair climbing, and squatting. Each item is assigned a weighted point value, and the total score ranges from 0 to 100, with higher scores indicating better knee function. Scores are commonly interpreted as: 95-100 excellent, 84-94 good, 65-83 fair, and <65 poor.

SECONDARY OUTCOMES:
MCID achievement rate | Preoperative, and 6 weeks, 3 months, 6 months, 12 months postoperatively
  Minimal Clinically Important Difference (MCID) achievement rate :
  1. For the target outcome, compute each participant's change from baseline to follow-up, signed so that improvement is positive (e.g., Δᵢ = Follow-up - Baseline for "higher=better"; Δᵢ = Baseline - Follow-up for "higher=worse").
  2. Mark a responder if Δᵢ ≥ MCID (or if using percent MCID: Δ%ᵢ = Δᵢ / Baseline × 100 ≥ MCID%).
  3. MCID achievement rate (%) = (number of responders ÷ number analyzed at that time point) × 100.
Operative time | Intraoperative
  Operative time is calculated as the interval from the first skin incision to completion of skin closure, recorded in minutes from the operating-room record.
Number of fluoroscopic shots | Intraoperative
  The total count of discrete single-image X-ray exposures acquired on the patient from first skin incision to completion of skin closure, as recorded by the C-arm exposure log/PACS.
Reoperation rate | 12 months postoperatively
  The proportion of patients requiring reoperation within 12 months of follow-up due to mechanical failure, fracture, or implant-related issues

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, M.D., Ph.D., Study Director — Department of Orthopaedic Surgery The First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
No IPD sharing is planned due to the high re-identification risk from radiographs/CT/MRI and 3D gait waveforms under our institution's privacy policy.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT07284524/Prot_SAP_000.pdf